CLINICAL TRIAL: NCT00798317
Title: A Randomized, Placebo Controlled, Double-masked, Multicenter Trial of Microplasmin Intravitreal Injection for Non-surgical Treatment of Focal Vitreomacular Adhesion.
Brief Title: Trial of Microplasmin Intravitreal Injection for Non-Surgical Treatment of Focal Vitreomacular Adhesion. The MIVI-TRUST (TG-MV-007) Trial.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-MV-007
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Vitreomacular Adhesion
MeSH Terms: interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ocriplasmin 125µg (Experimental): 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: Ocriplasmin 125µg
- Placebo (Placebo Comparator): Intravitreal injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocriplasmin 125µg — 125µg of ocriplasmin intravitreal injection
  Other Names: Microplasmin
  Arms: Ocriplasmin 125µg
Drug: Placebo — Intravitreal injection placebo.
  Arms: Placebo

SUMMARY:
This trial will evaluate the safety and efficacy of microplasmin, administered as an intravitreal injection, in subjects with focal vitreomacular adhesion. In previously performed clinical trials, some patients treated with intravitreal microplasmin have had resolution of their underlying condition, including macular hole closure, without need for vitrectomy. This clinical trial is justified because the sponsor believes the potential benefits outweigh the potential risks.

ELIGIBILITY:
Inclusion Criteria:

* Presence of focal vitreomacular adhesion (i.e., central vitreal adhesion within 6 mm Optical Coherence Tomography (OCT) field surrounded by elevation of the posterior vitreous cortex) that in the opinion of the Investigator is related to decreased visual function (such as metamorphopsia, decreased visual acuity, or other visual complaint)

Exclusion Criteria:

* Any evidence of proliferative retinopathy (including Proliferative Diabetic Retinopathy (PDR)) or other ischemic retinopathies involving vitreoretinal vascular proliferation) or exudative Age-Related Macular Degeneration (AMD) or retinal vein occlusion in the study eye
* Subjects with any vitreous hemorrhage or any other vitreous opacification which precludes either of the following: visualization of the posterior pole by visual inspection OR adequate assessment of the macula by either OCT and/or fluorescein angiogram in the study eye
* Subjects with macular hole diameter > 400 µm in the study eye
* Aphakia in the study eye
* High myopia (more than 8D) in study eye (unless prior cataract extraction or refractive surgery that makes refraction assessment unreliable for myopia severity approximation, in which case axial length >28 mm is an exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (20):
  - Retinal Diagnostic Center, Campbell, California
  - West Coast Retina Group, Inc, San Francisco, California
  - California Retina Consultants, Santa Barbara, California
  - Medeye, Miami, Florida
  - Retina Specialists, Pensacola, Florida
  - Paducah Retinal Center, Paducah, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Vision Research Center at Truman Medical Center, Kansas City, Missouri
  - Deleware Valley Retina Associates, Lawrenceville, New Jersey
  - Capital Region Retina, Albany, New York
  - Southeast Clinical Research Assoicates, PA, Charlotte, North Carolina
  - Dean A McGee Eye Institute, Oklahoma City, Oklahoma
  - Scheie Eye Institute, Penn Eye Care, Philadelphia, Pennsylvania
  - Black Hils regional Eye Institute, Rapid City, South Dakota
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants, Fort Worth, Texas
  - Medical Center Ophthalmology Assoc., San Antonio, Texas
  - Eye Care Associates, Tyler, Texas
  - Vitreoretinal Associates, Seattle, Washington
- University Hospital Leuven, Leuven, Belgium
- Czechia (6):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Kralovske Vinohrady, Prague
  - Central Military Hospital, Prague
  - Gemini Eye Clinic, Zlín
- Germany (10):
  - Augenklinik-Universität Bonn, Bonn
  - St. Joseph Stift Bremen Abteilung für Augenheilkunde, Bremen
  - Universitäts-Augenklinik Frankfurt am Main, Frankfurt
  - Städtische Kliniken Frankfurt am Main, Klinik für Augenheilkunde, Frankfurt am Main
  - Universität Göttingen, Göttingen
  - Klinik und Poliklinik für Augenheilkunde, Leipzig
  - Philipps Universität Marburg, Marburg
  - Augenklinik der Ludwig Maximilians Universität München, München
  - Augenärzte am St. Franziskus Hospital, Münster
  - Augenklinik im Dietrich-, Neubrandenburg
- Poland (2):
  - Indywidualna Specjalistyczna Praktyka Prywatna, Gdansk
  - Oddział Okulistyczny OSK,, Katowice
- Spain (5):
  - Instituto Oftalmología de Alicante (Vissum), Alicante
  - Centro Teknon-Institut de la Macula i de la Retina, Barcelona
  - Hospital La Paz, Madrid
  - Instituto Technologico de Oftalmologia S.L, Santiago de Compostela
  - Hospital General de Valencia, Valencia
- United Kingdom (4):
  - St Paul's Eye Unit, Liverpool
  - Moorfields Eye Hospital, London
  - Southampton Eye Unit, Southampton General Hospital, Southampton
  - Wolverhampton Eye Infirmary-New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Varma R, Haller JA, Kaiser PK. Improvement in Patient-Reported Visual Function After Ocriplasmin for Vitreomacular Adhesion: Results of the Microplasmin for Intravitreous Injection-Traction Release Without Surgical Treatment (MIVI-TRUST) Trials. JAMA Ophthalmol. 2015 Sep;133(9):997-1004. doi: 10.1001/jamaophthalmol.2015.1746. PMID 26068086
- [Derived] Folgar FA, Toth CA, DeCroos FC, Girach A, Pakola S, Jaffe GJ. Assessment of retinal morphology with spectral and time domain OCT in the phase III trials of enzymatic vitreolysis. Invest Ophthalmol Vis Sci. 2012 Oct 25;53(11):7395-401. doi: 10.1167/iovs.12-10379. PMID 23033391
- [Derived] Stalmans P, Benz MS, Gandorfer A, Kampik A, Girach A, Pakola S, Haller JA; MIVI-TRUST Study Group. Enzymatic vitreolysis with ocriplasmin for vitreomacular traction and macular holes. N Engl J Med. 2012 Aug 16;367(7):606-15. doi: 10.1056/NEJMoa1110823. PMID 22894573
- [Derived] DeCroos FC, Toth CA, Folgar FA, Pakola S, Stinnett SS, Heydary CS, Burns R, Jaffe GJ. Characterization of vitreoretinal interface disorders using OCT in the interventional phase 3 trials of ocriplasmin. Invest Ophthalmol Vis Sci. 2012 Sep 21;53(10):6504-11. doi: 10.1167/iovs.12-10370. PMID 22879421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was recruited on 23 Dec 2008 and last patient completed the study on 15 Jun 2010
Groups:
- Ocriplasmin 125µg: 125µg ocriplasmin intravitreal injection.
Period: Overall Study
Arm/Group | Ocriplasmin 125µg | Placebo
Started | 245 | 81
Completed | 235 | 74
Not Completed | 10 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin 125µg | Placebo | Total
Number analyzed (Participants) | 245 | 81 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (7.56) | 70.2 (10.85) | 72.0 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 56 | 222
  Male | 79 | 25 | 104

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Nonsurgical Resolution of Focal Vitreomacular Adhesion at Day 28
Description: Proportion of subjects with nonsurgical resolution of focal vitreomacular adhesion at Day 28, as determined by masked Central Reading Centre (CRC) Optical Coherence Tomography(OCT)evaluation.
Time Frame: Day 28
Population: Intention-To-Treat (ITT), Last Observation Carried Forward LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 125µg | Placebo
Number analyzed (Participants) | 245 | 81
percentage of participants | 25.3 | 6.2
Statistical Analysis 1: Comparison: Ocriplasmin 125µg vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — Comparing placebo and ocriplasmin; Odds Ratio (OR) = 5.13, 95% CI 2-sided [1.97 to 17.00]

2. Secondary Outcome: Proportion of Subjects With Total Posterior Vitreous Detachment (PVD) at Day 28
Description: Proportion of subjects with total PVD at Day 28, as determined by masked investigator assessment of B-scan ultrasound.
Time Frame: Day 28
Population: Intention-To-Treat (ITT), Last Observation Carried Forward LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 125µg | Placebo
Number analyzed (Participants) | 245 | 81
percentage of participants | 10.6 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs)/Serious Adverse Events (SAEs) were collected from injection day up to 6 months after injection
Description: AEs/SAEs were assessed by the investigator at all study visits
Groups:
- Ocriplasmin 125ug: 125ug ocriplasmin intravitreal injection
Arm/Group | Ocriplasmin 125ug | Placebo
Serious Adverse Events (participants affected / at risk) | 33/245 | 11/81
Other Adverse Events (participants affected / at risk) | 105/245 | 22/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 125ug (N=245) | Placebo (N=81)
Macular hole (Eye disorders) | 9 (9) | 5 (5)
Vitreous adhesions (Eye disorders) | 3 (3) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Hyphaema (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Eye disorders) | 1 (1) | 0 (0)
Wrist fracture (Eye disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Eye disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronay artery (Eye disorders) | 1 (1) | 0 (0)
Atrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal haemorrahge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Penumonia (Infections and infestations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Reumathoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 125ug (N=245) | Placebo (N=81)
Vitreous floaters (Eye disorders) | 38 (40) | 6 (8)
Conjuctival haemorrahge (Eye disorders) | 34 (34) | 10 (10)
Eye pain (Eye disorders) | 30 (33) | 5 (5)
Photopsia (Eye disorders) | 19 (21) | 1 (1)
Vision blurred (Eye disorders) | 17 (18) | 3 (3)
Visual acuity reduced (Eye disorders) | 13 (13) | 2 (2)
Macular oedema (Eye disorders) | 13 (13) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Varying agreements. The most restrictive is as follows: The Centre and Investigator agree to neither publish nor make public any of the results of the Study without the prior written consent from Sponsor, which consent shall not be unreasonably withheld.